CLINICAL TRIAL: NCT01755299
Title: Efficacy of "5-hour Energy"®, "5-Hour Energy Decaf"®, and Caffeine for Perceived Energy and Wakefulness
Brief Title: Efficacy of Energy Shots and Caffeine for Energy and Wakefulness Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProMedica Health System (Other)
Responsible Party: Principal Investigator, Michelle Piel, Pharmacy Resident, ProMedica Health System
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 5HE-TOL
Record Dates: First submitted 2012-12-18; First posted 2012-12-24 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Focus: to Compare a Commercially Available Energy Drink, B Vitamins, Caffeine Alone, and Placebo for Effectiveness on Perceived Energy Level and Wakefulness
Keywords: Energy drinks; Wakefulness; Caffeine
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Active ingredient (Active Comparator): Regular "5-hour Energy"
  Interventions: Other: Regular "5-hour Energy"
- Active ingredient-2 (Active Comparator): "5-hour Energy Decaf"
  Interventions: Other: Decaf "5-hour Energy"
- Active ingredient-3 (Active Comparator): Compounded caffeine product 135 mg/2 ounces
  Interventions: Other: Compounded concentrated caffeine liquid
- Placebo (Placebo Comparator): Flavored placebo
  Interventions: Other: Flavored bottled water

INTERVENTIONS:
Other: Regular "5-hour Energy" — Amount equivalent to the package commercially packaged and sold (1.93 fl. oz.)
  Other Names: Original brand "5-Hour Energy" product
  Arms: Active ingredient
Other: Decaf "5-hour Energy" — Commercially available "5-Hour Energy Decaf" product in the amount that is packaged (1.93 fl. oz.)
  Other Names: "5-hour Energy Decaf"
  Arms: Active ingredient-2
Other: Compounded concentrated caffeine liquid — Concentrated caffeine liquid has been used to compound a 135 mg/2 ounce caffeine product, which contains the same amount of caffeine as a regular "5-hour Energy"
  Arms: Active ingredient-3
Other: Flavored bottled water — Bottled water will be flavored and colored to serve as a placebo product for this trial.
  Other Names: Water; Placebo
  Arms: Placebo

SUMMARY:
The line of "5-hour Energy"® products are available over-the-counter as energy supplements. The appeal of these products involves ease of use, low caloric value, and the absence of sugar to prevent a "crash" later in the day. The definitive efficacy and potency of the products is unknown due to the lack of evidence-based clinical reports. It is suspected that the efficacy related to these products is due to the caffeine content, which was reported as 138 mg per 2-ounce bottle in an online caffeine content chart. The purpose of this randomized, double-blind, placebo controlled, four way crossover study is to evaluate the efficacy of "5-hour Energy"®, "5-Hour Energy Decaf"®, caffeine, and placebo for perceived energy and wakefulness.

DETAILED DESCRIPTION:
Please see brief summary contained above.

ELIGIBILITY:
Inclusion Criteria: Subjects must be age 18 years or older who consume no more than five caffeinated beverages and products per day. One caffeinated beverage is defined as any of the following: six ounces of cold or hot coffee or tea, twelve ounces of soda with caffeine, or one energy drink.

Exclusion Criteria:

* Age less than 18 years
* Subjects who are pregnant or breast-feeding
* Diagnosis of any of the following disease states:

  * Attention Deficit Hyperactive Disorder
  * Anxiety
  * Coronary Artery Disease
  * Cardiac arrhythmias
  * Cerebral vascular accident
  * Narcolepsy
  * Seizure disorders
  * Uncontrolled hypertension
* Active therapy with stimulant medications - any medications containing amphetamine, atomoxetine, dextroamphetamine, diethylpropion, lisdexamfetamine, methylphenidate, phentermine, or modafinil
* Use of decongestants or other products containing phenylephrine or pseudoephedrine for more than 15 days within the past 30 days
* Subjects who work third shift or rotate to two or more different shifts for their job, not allowing them to have a regular sleep schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Subjective wakefulness levels based on assessment tool rankings | At one, three, and five hours after taking the study product
  Subjects are provided with assessment tools to use for each product. The tool contains the Stanford Sleepiness Scale to assess for wakefulness levels. All appropriate options are listed, and subjects are required to circle one option at one, three, and five hours after taking the study product for the day.

SECONDARY OUTCOMES:
Number of patients experiencing adverse effects associated with study products | Within five hours after taking study product
  Each assessment tool has a space for subjects to list any side effects that were experienced throughout the five hour period of time after taking a study product.

OTHER OUTCOMES:
Study product consumed | Within the five hours after taking the study product
  There is a space on each assessment tool for patients to guess what study product they think that they consumed on that date.

CONTACTS AND LOCATIONS:
Locations (1):
- Flower Hospital Family Medicine Residency, Sylvania, Ohio, United States

REFERENCES:
- See also: Energy Shots Review — http://www.webmd.com/food-recipes/features/energy-shots-review
- See also: 5-hour Energy Website — http://www.5hourenergy.com
- See also: Source for caffeine content of many commercially available products — http://www.energyfiend.com/the-caffeine-database